CLINICAL TRIAL: NCT03596554
Title: X-linked Hypophosphatemia and Carbohydrate and Lipid Metabolism: a Role for FGF21?
Brief Title: X-linked Hypophosphatemia and FGF21
Acronym: XLH 21
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0349; 2018-A01304-51 (Other: ID-RCB)
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: X-linked Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Descriptive study — Description of the circulating values of Fibroblast Growth Factor 21 in X-linked hypophosphatemia children compared to controls in the VITADOS cohort (healthy children and adolescents aged 10-18 years), after age-matched, pubertal stage and sex).

SUMMARY:
Fibroblast Growth Factor 23 and Fibroblast Growth Factor 21 are two endocrine Fibroblast Growth Factors, requiring Klotho as a co-factor to promote their systemic actions. Fibroblast Growth Factor 21 is involved in the regulation of glucid and lipid metabolism. Fibroblast Growth Factor 21 Knock Out mice display obesity and hyperglycemia.

In investigators experience, patients with X-linked hypophosphatemia often present with early-onset over-weight that could be partly explained by decreased physical activity because of bone pains and deformations after puberty; however, patients usually display progressive over-weight earlier in life, when there is no limitation of physical activity yet.

To the knowledge of investigators the association between Fibroblast Growth Factor 23, Fibroblast Growth Factor 21 and Klotho in patients with X-linked hypophosphatemia has never been evaluated. Thus, the main objective of this study is to evaluate the glucid and lipid metabolism in patients with X-linked hypophosphatemia, the main working hypothesis being that the genetic deregulation in the Fibroblast Growth Factor 23 axis in patients with X-linked hypophosphatemia induces modifications of Klotho levels (namely decreased levels) that in turn will deregulate the Fibroblast Growth Factor 21 axis (resistance to Fibroblast Growth Factor 21 because of decreased Klotho levels).

ELIGIBILITY:
Inclusion Criteria:

* Child with X-linked hypophosphatemia with PHEX gene mutation
* Child between 10 and 18 years old
* Child over 10 kg having a blood sample as part of the treatment (due to regulatory constraints for blood volume taken in 30-day period of 40 mL in children over 10 kg)
* Child and parent / holder of parental authority who has been informed of the study and does not object to participate.

Exclusion Criteria:

- Pregnancy in progress

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients aged 10 to 18 years followed in the different sites of the French Reference Center for Rare Diseases of Calcium and Phosphate, and monitored for hypophosphatemic rickets; estimated number to be included, N=40
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Circulating FGF21 | 1 day
  Samples specific to the study will be collected during a sampling performed as part of the usual care and follow-up of the patient. An additional tube (5 ml maximum) will be collected, which will be sent to the Lyon Sud Hospital Center for analysis of circulating FGF21.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre de Référence des Maladies Rénales Rares - Centre de Référence des Maladies Rares du Calcium et du Phosphate - Service de Néphrologie, Rhumatologie et Dermatologie Pédiatriques - Hôpital Femme Mère Enfant, Bron
  - Centre de Référence des Maladies Rares du Calcium et du Phosphore, Service d'Endocrinologie Pédiatrique - Hôpital du Kremlin Bicêtre, Paris
  - Endocrinologie, Maladies Osseuses, Gynécologie, Génétique, Hôpital des Enfants, CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No